CLINICAL TRIAL: NCT02656433
Title: Transcranial Noninvasive Brain Stimulation With Random Noise for Children With Congenital or Acquired Brain Injury
Brief Title: tES With Random Noise Stimulation Applied to Children With Brain Injury
Acronym: BrainInjury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRNS23062015
Record Dates: First submitted 2015-11-21; First posted 2016-01-15 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Brain Injury; Motor Skills Disorders
Keywords: QEEG; ERP; tRNS; Brain injury; Motor Impairment; Transcranial Brain non-invasive stimulation; electroencephalogram
MeSH Terms: conditions — Brain Injuries; Motor Skills Disorders | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Receive treatment with physiotherapy
  Interventions: Other: Physiotherapy
- Experimental or tRNS Group (Experimental): Receive treatment with physiotherapy plus Transcranial Random Noise Stimulation (tRNS)
  Interventions: Device: Transcranial Random Noise Stimulation; Other: Physiotherapy

INTERVENTIONS:
Device: Transcranial Random Noise Stimulation — A special Helmet supply weak electrical currents in the head
  Other Names: tRNS
  Arms: Experimental or tRNS Group
Other: Physiotherapy — Standard of care physiotherapy aimed to the motor impairment the subject presents

SUMMARY:
50 children between 4 and 7 years old with moderate to severe motor impairment, 50% males 50% females will participate in an interventional study in two groups: placebo and experimental group.

Placebo group will only receive traditional treatment with physiotherapy and the Experimental or tRNS Group will receive physiotherapy plus tRNS BrainNoninvasive Stimulation.

DETAILED DESCRIPTION:
In this Interventional Study with Double Blind Assignment to Placebo and Experimental Group, Gross Motor Function Measure (GMFM) and Neurophysiological are the parameters measured with EEG amplifier before and after 30 sessions.

Work hypothesis is that the tRNS Group will present better motor functionality after 30 sessions of 30 minutes of duration of electrical brain stimulation administered during physiotherapy exercises 2 days per week than the Group that only receives treatment with physiotherapy during 30 minutes 2 days per week without tRNS.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 3 and 7 years.
* Meet criteria for Congenital or Acquired Brain Injury .
* Patients who have been diagnosed at least 1 year before inclusion in the study.

Exclusion Criteria:

* Acute visual or hearing loss.
* Other neurological disorders: migraine, epilepsy, tuberous sclerosis
* Other neurodevelopmental disorders like ASD, ADHD, PDD, etc ...

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) as measured by the Gross Motor Function scale | Up to five months
  Motor Functionality Scale

SECONDARY OUTCOMES:
Differences in Power Fast Fourier Transformation before and after intervention | up to five months
  Changes in Power in EEG over different electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Moises Aguilar Domingo, PhD, Principal Investigator — Fundación Española para el Desarrollo de la Neurometria (Brainmech)
Locations (1):
- New Remedies, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Bashir S, Yoo WK. Cheap Technology Like Transcrinal Direct Current Stimulation (tDCS) Could Help in Stroke Rehabilitation in South Asia. Basic Clin Neurosci. 2013 Summer;4(3):188-9. No abstract available. PMID 25337347
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Result] Benninger DH, Lomarev M, Lopez G, Wassermann EM, Li X, Considine E, Hallett M. Transcranial direct current stimulation for the treatment of Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Oct;81(10):1105-11. doi: 10.1136/jnnp.2009.202556. PMID 20870863
- [Result] Fregni F, Boggio PS, Valle AC, Rocha RR, Duarte J, Ferreira MJ, Wagner T, Fecteau S, Rigonatti SP, Riberto M, Freedman SD, Pascual-Leone A. A sham-controlled trial of a 5-day course of repetitive transcranial magnetic stimulation of the unaffected hemisphere in stroke patients. Stroke. 2006 Aug;37(8):2115-22. doi: 10.1161/01.STR.0000231390.58967.6b. Epub 2006 Jun 29. PMID 16809569
- [Result] Vanneste S, Fregni F, De Ridder D. Head-to-Head Comparison of Transcranial Random Noise Stimulation, Transcranial AC Stimulation, and Transcranial DC Stimulation for Tinnitus. Front Psychiatry. 2013 Dec 18;4:158. doi: 10.3389/fpsyt.2013.00158. eCollection 2013. PMID 24391599
- [Result] Fregni F, Otachi PT, Do Valle A, Boggio PS, Thut G, Rigonatti SP, Pascual-Leone A, Valente KD. A randomized clinical trial of repetitive transcranial magnetic stimulation in patients with refractory epilepsy. Ann Neurol. 2006 Oct;60(4):447-55. doi: 10.1002/ana.20950. PMID 17068786
- [Result] Fertonani A, Pirulli C, Miniussi C. Random noise stimulation improves neuroplasticity in perceptual learning. J Neurosci. 2011 Oct 26;31(43):15416-23. doi: 10.1523/JNEUROSCI.2002-11.2011. PMID 22031888
- [Result] Ilyukhina VA, Kozhushko NY, Matveev YK, Ponomareva EA, Chernysheva EM, Shaptilei MA. Transcranial micropolarization in the combined therapy of speech and general psychomotor retardation in children of late preschool age. Neurosci Behav Physiol. 2005 Nov;35(9):969-76. doi: 10.1007/s11055-005-0153-7. PMID 16270180
- [Result] McCleery JP, Elliott NA, Sampanis DS, Stefanidou CA. Motor development and motor resonance difficulties in autism: relevance to early intervention for language and communication skills. Front Integr Neurosci. 2013 Apr 24;7:30. doi: 10.3389/fnint.2013.00030. eCollection 2013. PMID 23630476
- [Result] Mueller A, Candrian G, Kropotov JD, Ponomarev VA, Baschera GM. Classification of ADHD patients on the basis of independent ERP components using a machine learning system. Nonlinear Biomed Phys. 2010 Jun 3;4 Suppl 1(Suppl 1):S1. doi: 10.1186/1753-4631-4-S1-S1. PMID 20522259
- [Result] Mueller A, Candrian G, Grane VA, Kropotov JD, Ponomarev VA, Baschera GM. Discriminating between ADHD adults and controls using independent ERP components and a support vector machine: a validation study. Nonlinear Biomed Phys. 2011 Jul 19;5:5. doi: 10.1186/1753-4631-5-5. PMID 21771289
- [Result] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Result] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Result] Nitsche MA, Nitsche MS, Klein CC, Tergau F, Rothwell JC, Paulus W. Level of action of cathodal DC polarisation induced inhibition of the human motor cortex. Clin Neurophysiol. 2003 Apr;114(4):600-4. doi: 10.1016/s1388-2457(02)00412-1. PMID 12686268
- [Result] Nitsche MA, Doemkes S, Karakose T, Antal A, Liebetanz D, Lang N, Tergau F, Paulus W. Shaping the effects of transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2007 Apr;97(4):3109-17. doi: 10.1152/jn.01312.2006. Epub 2007 Jan 24. PMID 17251360
- [Result] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Result] Paulus W. Transcranial electrical stimulation (tES - tDCS; tRNS, tACS) methods. Neuropsychol Rehabil. 2011 Oct;21(5):602-17. doi: 10.1080/09602011.2011.557292. Epub 2011 Aug 5. PMID 21819181
- [Result] Priori A, Berardelli A, Rona S, Accornero N, Manfredi M. Polarization of the human motor cortex through the scalp. Neuroreport. 1998 Jul 13;9(10):2257-60. doi: 10.1097/00001756-199807130-00020. PMID 9694210
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Result] Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. Arch Neurol. 2008 Dec;65(12):1571-6. doi: 10.1001/archneur.65.12.1571. PMID 19064743
- [Result] Schneider HD, Hopp JP. The use of the Bilingual Aphasia Test for assessment and transcranial direct current stimulation to modulate language acquisition in minimally verbal children with autism. Clin Linguist Phon. 2011 Jun;25(6-7):640-54. doi: 10.3109/02699206.2011.570852. Epub 2011 Jun 1. PMID 21631313
- [Result] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- See also: Neurometrics — http://www.neurometrics.es